CLINICAL TRIAL: NCT03564925
Title: Comparison of Wide Area Circumferential Ablation With Cryoballoon Ablation in Patients With Paroxysmal Atrial Fibrillation: A Multi-center, Prospective, Randomized, Controlled Study
Brief Title: Wide Area Circumferential Ablation With Contact Force Versus Cryoballoon Ablation
Acronym: WACACF vs Cryo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Proffessor, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WACACF vs Cryo
Record Dates: First submitted 2017-09-10; First posted 2018-06-21 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation; CryoAblation; Pulmonary Vein Isolation
Keywords: Atrial Fibrillation; CryoAblation; pulmonary vein isolation; wide area circumferential ablation; contact force
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: two groups, group one is for Wide Area Circumferential Ablation With Contact Force catheter, group two is for Cryoballoon Ablation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wide area circumferential ablation (Active Comparator): Device:Smart Touch® Irrigated Tip Ablation Catheter in combination with 3D mapping system CARTO or any future development generations of this product line, provided they are CE marked and the centre has the experience of at least 10 procedures before including a patient into the study.
  Interventions: Procedure: Wide area circumferential ablation
- Cryoballoon ablation (Experimental): Device: ArcticFront® Cardiac CryoAblation Catheter System with the FlexCath Steerable Sheath or ArcticFront® Advance Cardiac CryoAblation Catheter System with the FlexCath Steerable Sheath or any future development generations of this product line, provided they are CE marked and the centre has the experience of at least 10 procedures before including a patient into the study.
  Interventions: Procedure: Cryoballoon ablation

INTERVENTIONS:
Procedure: Wide area circumferential ablation — Wide area circumferential ablation with contact force catheter will be performed in Patients allocated in this group,the induction of atrial fibrillation by isoproterenol or programmed stimulation and burst pacing will be performed. If frequent atrial premature beats are found beyond pulmonary vein, activation mapping will be performed for eliminating the triggers. If atrial tachycardias(ATs)are induced, activation mapping the ATs and ablation will be performed. Electrical isolation of pulmonary veins and elimination the triggers and ATs induced by isoproterenol or programmed stimulation and burst pacing are the endpoints of ablation
  Arms: Wide area circumferential ablation
Procedure: Cryoballoon ablation — In the cryoballoon procedures, pulmonary vein isolation (PVI) was achieved using fluoroscopic guidance to position the cryoballoon catheter. Once PV-to-balloon occlusion was confirmed by retrograde radiopaque contrast agent retention, circumferential ablation was performed by freezing with a single-shot delivery of coolant to the balloon.
  Arms: Cryoballoon ablation

SUMMARY:
The purpose of this randomized clinical trial is to compare the efficacy and safety of wide area circumferential ablation using contact force catheter with cryoballoon ablation for the treatment of paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and is associated with stroke, reductions in quality of life and overall survival. Previous studies have shown that cryoballoon ablation was noninferior to radiofrequency ablation with respect to efficacy for the treatment of patients with drug-refractory paroxysmal atrial fibrillation. However, the pulmonary vein isolation for radiofrequency catheter ablation in previous studies was done around each pulmonary-vein antrum, and it's not wide area circumferential ablation. Moreover, the induction of atrial fibrillation by isoproterenol or programmed stimulation and burst pacing was not performed in most of previous studies. We hypothesize that wide area circumferential ablation with contact force catheter and combined catheter ablation the potential atrial triggers and/or other atrial arrhythmias induced by aggressive induction is more effective than cryoballoon ablation in patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic PAF with at least two episodes and at least one episode documented (30 seconds episode length, documented by ECG within last 12 months).

   Documented treatment failure for effectiveness of at least one anti-arrhythmic drug(AAD Type I or III, including β-blocker and AAD intolerance).
2. ≥ 18 and ≤ 75 years of age.
3. Patients who are mentally and linguistically able to understand the aim of the trial and to show sufficient compliance in following the trial protocol.
4. Patient is able to verbally acknowledge and understand the associated risks, benefits, and treatment alternatives to therapeutic options of this trial: cryoballoon ablation system or standard RF ablation technique. The patients, by providing informed consent, agree to these risks and benefits as stated in the patient informed consent document. All the details have been presented to him and he has signed the informed consent form for the trial.

Exclusion Criteria:

Exclusion criteria related to a cardiac condition

1. Patients with prosthetic valves.
2. Any previous LA ablation or surgery.
3. Any cardiac surgery or percutaneous coronary intervention (PCI) within three months prior to enrollment.
4. Unstable angina pectoris.
5. Myocardial infarction within three months prior to enrollment.
6. Symptomatic carotid stenosis.
7. Chronic obstructive pulmonary disease with detected pulmonary hypertension.
8. Any condition contraindicating chronic anticoagulation.
9. Stroke or transient ischemic attack within six months prior to enrollment.
10. Any significant congenital heart defect corrected or not (including atrial septal defects or PV abnormalities) but not including patent foramen ovale.
11. New York Heart Association (NYHA) class III or IV congestive heart failure.
12. EF < 35 % (determined by echocardiography within 60 days of enrollment as documented in patient medical history).
13. Anteroposterior LA diameter > 55 mm (by trans-thoracic echocardiography (TTE or TEE) within three months to prior enrollment).
14. LA thrombus (TEE diagnostic performed on admission). Intracardiac thrombus.
15. PV diameter > 26 mm in right sided PVs.
16. Mitral prosthesis.
17. Hypertrophic cardiomyopathy
18. 2° (Type II) or 3° atrioventricular block.
19. Brugada syndrome or long QT syndrome.
20. Arrhythmogenic right ventricular dysplasia.
21. Sarcoidosis.
22. PV stent.
23. Myxoma.

Exclusion criteria based on laboratory abnormalities

1. Thrombocytosis (platelet count > 600,000 / µl), thrombocytopenia (platelet count < 100,000 / µl).
2. Any untreated or uncontrolled hyperthyroidism or hypothyroidism.
3. Severe renal dysfunction (stage V, requiring or almost requiring dialysis, glomerular filtration rate (GFR) < 15 ml / min).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to first documented recurrence of atrial arrhythmias | 12 months
  a blanking period of three months will be maintained after the initial procedure

SECONDARY OUTCOMES:
time to the first occurrence of each of the components of the primary outcome | 12 months
  a blanking period of three months will be maintained after the initial procedure
all-cause death | 12 months
  all-cause death
Arrhythmia-related death | 12 months
  Arrhythmia-related death
total procedural duration | 12 months
  time of total procedural
total time of fluoroscopy | 12 months
  total time of fluoroscopy
time to recurrent atrial fibrillation (AF) | 12 months
  a blanking period of three months will be maintained after the initial procedure
time to first cardiovascular hospitalization | 12 months
  a blanking period of three months will be maintained after the initial procedure
number of cardiovascular hospitalizations (over-night stays) | 12 months
  a blanking period of three months will be maintained after the initial procedure
quality of life changes at 12 months compared to baseline | 12 months
  with the evaluation of the MOS item short from health survey（SF-36）
time to first symptomatic AF recurrence | 12 months
  a blanking period of three months will be maintained after the initial procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affilliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964